CLINICAL TRIAL: NCT00347711
Title: Bevacizumab and Retinal Vascular Occlusions
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: APEC-0020
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Edema Macular; Vascular Occlusion
MeSH Terms: conditions — Macular Edema | interventions — Intravitreal Injections

INTERVENTIONS:
Drug: Intravitreal injection

SUMMARY:
To evaluate the effects of Intravitreal Bevacizumab in macular edema in retinal vascular occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Vascular occlusion and edema macular diagnosticated by fluorescein angiography and coherent optic tomography

Exclusion Criteria:

* Previous surgery
* Uveitis
* Glaucoma

Ages: 40 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Griselda Alvarez, Fellow, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociacion para Evitar la Ceguera en Mexico, México, D.F. Mexico, Mexico